CLINICAL TRIAL: NCT01176643
Title: Development and Evaluation of an Adapted Yoga Program as Adjunct Therapy for Persons With Systemic Lupus Erythematosus (SLE): a Pilot Study
Brief Title: Development and Evaluation of Modified Yoga in Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Sasha Bernatsky, DR, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GEN10-037
Record Dates: First submitted 2010-07-30; First posted 2010-08-06 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Yoga
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Standard of Care; Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard care plus yoga (Active Comparator): Participants will be asked to complete two yoga classes weekly over a period of eight weeks.
  Interventions: Other: Standard care plus Yoga
- Standard care (No Intervention)

INTERVENTIONS:
Other: Standard care plus Yoga — Participants will be asked to complete two yoga classes weekly over a period of eight weeks.
  Arms: standard care plus yoga

SUMMARY:
The purpose of this study is to test the effects of a modified yoga program in persons with SLE.

DETAILED DESCRIPTION:
Background and relevance: Systemic lupus erythematosus (SLE) is an autoimmune disease characterized by multisystem inflammation that leads to numerous clinical manifestations which can potentially result in permanent organ damage. In Canada, it is estimated that 1 woman in every 2000 has SLE, with peak incidence occurring in women of childbearing age. Although survival rate has improved, physical and psychological health status remains significantly impaired. With its increasing prevalence, its morbidity, and the complexities associated with side effects related to its treatment, SLE presents a treatment challenge to the clinician. Nonpharmacological interventions that incorporate holistic, mind-body, approaches aimed at improving physical and psychological health in persons with SLE are needed.

Recent studies have shown a number of physical and mental health benefits associated with yoga among persons with various chronic conditions. In SLE, no study has been undertaken to specifically tailor and evaluate the feasibility and potential benefits of a yoga program for this patient population. We developed a yoga program, based on Iyengar yoga, to address needs specific to persons with lupus, taking into account the physical and psychological effects of this illness.

Hypothesis: Persons with SLE will benefit from an adapted yoga program with improved health status including, decreased psychological distress, fatigue, pain, and improved physical conditioning and quality of life.

Objectives: To 1) develop a standardized yoga program adapted specifically to persons with SLE, 2) evaluate the feasibility of using the yoga program in SLE, and 3) determine the effect of the yoga program on psychological distress, fatigue, pain, physical conditioning, and overall quality of life in SLE.

Methodology: This will be a randomized control study. Participants will be recruited at the McGill University Health Centre Lupus Clinic. Consenting participants will be randomly allocated to standard treatment (control group) or standard treatment plus yoga (treatment group). We expect to recruit 24 persons in each group.

All participants will have physical assessments of disease activity and damage performed by their physician at study entry and at study completion. Questionnaires addressing psychological and physical distress will be administered at entry and at the completion of the study. Participants in the yoga group will be asked to attend 60-minute yoga classes twice weekly for a period of eight weeks. The classes will be held in a yoga studio and led by a certified Iyengar yoga instructor. The program consists of a series of poses. Focusing on correct body alignment, the instructor will lead participants into poses that concentrate on relaxing muscle to release physical tension and create mental relaxation. Props (blankets, bolsters, blocks) will be used to attain poses with ease. All poses will be taught with the intention that they will be easily replicated at home.

Expected outcome: It is expected that the yoga program will provide a valuable coping tool for managing SLE manifestations and improving physical and psychological distress caused by the symptoms and treatments of SLE.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* Diagnosis of SLE based on ACR criteria

Exclusion Criteria:

* presently enrolled in a yoga program
* osteoporosis (T score ≥ -2.5)
* avascular necrosis
* taking quinolone in the preceding 3 months
* taking ≥ 30 mg of prednisone daily
* history of joint replacement or organ transplant
* Persons with any pre-existing condition that would prevent attendance at the yoga classes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Measures of compliance (class attendance, frequency of home practice)and results of post-yoga evaluations and post yoga discussion groups will be used as measures of feasibility of using yoga in SLE | 3 months (post yoga intervention)
  The number of yoga classes attended and homework logs will be monitored. Post-yoga evaluations will be used to assess satisfaction, acceptability, feasibility and perceived helpfulness of the yoga program. Audiotaped discussion groups led by an experienced moderator will follow the last yoga class. Content analysis will be used to analyze recorded transcripts.

SECONDARY OUTCOMES:
Pre- and post-yoga measurements of disease activity, quality of life, psychological distress (depression,anxiety and stress), sleep quality, fatigue, pain, and a global assessment of health will be used to assess efficacy of yoga in SLE | 3 months (post yoga intervention)
  Disease activity will be assessed by a medical evaluator blinded to the study hypothesis at study entry and at completion of the yoga program. Self-report questionnaires will be used to measure pre- and post-yoga assessments of quality of life (SF36), psychological distress (CESD, STAI and PSS), sleep quality (PSQI),fatigue (MFI20),and visual analogue scales will be used to measure pain and self-reported health.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre at Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Badsha H, Chhabra V, Leibman C, Mofti A, Kong KO. The benefits of yoga for rheumatoid arthritis: results of a preliminary, structured 8-week program. Rheumatol Int. 2009 Oct;29(12):1417-21. doi: 10.1007/s00296-009-0871-1. Epub 2009 Jan 31. PMID 19184028